CLINICAL TRIAL: NCT04326868
Title: Human Soil Transmitted Helminths (STH) Resistance to Benzimidazole in School Aged Children Living in Gabon
Acronym: BenziR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre de Recherche Médicale de Lambaréné (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0084/2019/PR/SG/CNER; CEI- 007/2019 (Other: Institutional ethics committee)
Record Dates: First submitted 2020-03-04; First posted 2020-03-30 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Helminths Infection; Drug Resistance
Keywords: Helminths; Resistance; Gabon; Infection; CERMEL; Benzimidazole
MeSH Terms: conditions — Infections | interventions — Albendazole; Mebendazole; Pyrantel

STUDY DESIGN:
Intervention Model Description: The participants diagnosed positive for Soil Helminths Infection will be randomly assigned to one of the following treatment arms of the study.
  Parents or guardians of eligible children will be asked to bring them to the CERMEL (clinic). after a brief clinical examination child fulfilling inclusion criteria will be randomly assigned to one of the following treatment regimens of the study. These regimens consisted of treatment as follow: given as a single tablet once daily for 3 consecutive days
  * A single tablet of ABZ (400mg), administered during 3 consecutive days;
  * 1 tablet of ABZ 400mg + 1 tablet of MBZ (500mg) administered in 3 consecutive days,
  * 1 tablet of ABZ (400mg) + Pyr (125 mg) administered in 3 consecutive days
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Albendazole (Active Comparator): ABZ (400mg)
  Interventions: Drug: Benzimidazole Anthelmintic
- Albendazole and Mebendazole (Experimental): ABZ 400mg + 1 tablet of MBZ (500mg)
  Interventions: Drug: Benzimidazole Anthelmintic
- Albendazole and Pyrantel (Experimental): ABZ (400mg) + Pyr (125 mg)
  Interventions: Drug: Benzimidazole Anthelmintic

INTERVENTIONS:
Drug: Benzimidazole Anthelmintic — The participants diagnosed positive will be randomly assigned to one of the following treatment arms of the study. Parents or guardians of eligible children will be asked to bring them to the CERMEL (clinic). after a brief clinical examination child fulfilling inclusion criteria will be randomly assigned to one of the following treatment regimens of the study.
  Other Names: Albendazole; Mebendazole; Pyrantel

SUMMARY:
Soil-transmitted helminths (STHs) infections are common in subtropics and mostly affect the poorest communities, with an impact on human health in many parts of the world. In 2017, World Health organization (WHO) reports more than 1.5 billion people are infected with soil-transmitted helminths worldwide, including 568 million school-age children who need treatment and preventive interventions. Preventive chemotherapy and periodic mass administration with benzimidazoles (BZ) [albendazole (ABZ) and mebendazole (MBZ)] are used to control these parasites. However, rapid reinfection with Ascaris lumbricoides within six months after a completed treatment has been reported, while the reinfection with hookworms is slow. Similarly, the efficacy of these drugs on Trichuris trichiura cure rate is poor. After many years of use of this drug class, there is an increase possibility that BZ resistance could develop. This resistance may occur due to single nucleotide polymorphisms (SNPs) in the β-tubulin gene at positions 167, 198 or 200, as has been reported in animals. Little data exist to show whether any of these polymorphisms do influence the BZ efficacy against STH in humans. The present study will develop methods to look for molecular evidence of BZ drug resistance in human population in order to support the investigation of the control and elimination of neglected tropical diseases (NTDs) in our communities.

DETAILED DESCRIPTION:
A Randomized Controlled Clinical Trial (RCT) cohort study, to evaluate the efficacy and safety of three benzimidazole derivates drug (Albendazole, Mebendazole, Albendazole Mebendazole, and Albendazole-Pyrantel) to treat major STH in school aged children from Lambaréné and surroundings. After obtaining informed consent from parents or guardians, stool samples will be collected, for infectious status. If positive the participant will be treated with either drug combination. The efficacy and SNP frequencies will be assessed at weeks 3 and 6 post treatment

Description of study population Children of school and preschool age (2 to 17 years old) living in Lambaréné and the surrounding areas are eligible. The choice of school and preschool-aged children is based on the fact that they constitute the main population at risk of infection. In addition, most of the resources available for public health interventions in many endemic areas of soil-transmitted helminths target this group as a cost-effective method for reaching a large part of the population.

The previous analysis of patient cohort reported a success rate of 61% multispecies prevalence amongst children in the study area and considering a significance level of 95% confidence interval (α =5%) and a minimum power of 80%, the investigators will have to include a total of 255 participants in the study

ELIGIBILITY:
Inclusion Criteria:

* Living in Lambaréné and surrounding areas
* Written informed consent or assent
* Microscopy positive for any major Soil-Transmitted helminths

Exclusion Criteria:

* Microscopy negative for any STH
* Pregnant women
* Do not be available for followed up.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 255 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Assessment of eggs rate reduction . | three weeks to six weeks
  The assessment of efficacy will be the level of the eggs rate reduction . The assessment will be done at weeks 3 and 6 and a different treatment regimen will be compared according to protocol and intention to treat.
  This evaluation will be based on the same parasitological examinations carried out at the beginning. Using polymerase chain reaction(PCR) for a better, appreciation of the efficacy of Benzimidazole.
Assessment of cure rate | three weeks to six weeks
  The assessment of efficacy as a cure rate, based on the absence of eggs at three and six weeks post treatment, using microscopy and PRC examination.

SECONDARY OUTCOMES:
The assessment of safety | three to six weeks.
  The adverse events due to a drug intake and the frequency of single nucleotide polymorphisms (SNPs) before and after treatment in each group.The safety of administration of Benzimidazole will be evaluated primarily clinically. The safety will be evaluated within 24 hours and at any unscheduled visit or at week 3 and week 6 to record any symptoms that occur after the drug has been administered.

CONTACTS AND LOCATIONS:
Overall Officials: Ayôla Akim ADEGNIKA, Principal Investigator — Centre de Recherche Médicale de Lambaréné
Locations (1):
- Centre de Recherches Médicales de Lammbaréné, Lambaréné, Moyen-Ogooué Province, Gabon

IPD SHARING:
Plan to Share IPD: Yes
The Data will be shared in RedCap database.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The date will be available around December 2020 until september 2021.
Access Criteria: The Data will be shared12 months after study completion in research journal. A lle the result will be publicly available the

REFERENCES:
- [Derived] Nguema Moure PA, Nzamba Maloum M, Manouana GP, Laclong Lontchi R-A, Mbong Ngwese M, Edoa JR, Frejus Zinsou J, Meulah B, Mahmoudou S, N'noh Dansou EM, Josiane Honkpehedji Y, Romeo Adegbite B, Agnandji ST, Ramharter M, Lell B, Borrmann S, Kremsner PG, Dejon-Agobe JC, Adegnika AA. A randomized assessors-blind clinical trial to evaluate the safety and the efficacy of albendazole alone and in combination with mebendazole or pyrantel for the treatment of Trichuris trichiura infection in school-aged children in Lambarene and surroundings. Antimicrob Agents Chemother. 2024 May 2;68(5):e0121123. doi: 10.1128/aac.01211-23. Epub 2024 Apr 2. PMID 38563751